CLINICAL TRIAL: NCT06221735
Title: Evaluating the Accuracy of New Tests for TB Infection Diagnosis
Acronym: TB infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freundeskreis Für Internationale Tuberkulosehilfe e.V (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TBI Testing
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Latent Tuberculosis; TB Infection; Tuberculosis
Keywords: Tuberculosis; TB Infection; LTBI; TBI
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Intervention Model Description: Participants will be injected with Cy-TB and the results will be read after 48-72 hours. 10 mL of blood will be obtained from each participant and transferred to three TB-Feron tubes and four QFT-Plus tubes whereby the tubes will be incubated at 37℃ for 16 to 24 hours. The TB-Feron tubes will be analyzed with the fully automated STANDARD F2400 device, while QFT-Plus tubes will be analyzed using an ELISE microplate reader
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cy-TB test (Experimental): The study will include people with confirmed TB infection and negative controls to compare the specificity and sensitivity of the Cy-TB and TB-Feron tests versus the QFT-Plus assay
  Interventions: Diagnostic Test: Cy-TB test; Diagnostic Test: STANDARD F TB-Feron FIA test
- STANDARD F TB-Feron FIA test (Experimental): The study will include people with confirmed TB infection and negative controls to compare the specificity and sensitivity of the Cy-TB and TB-Feron tests versus the QFT-Plus assay
  Interventions: Diagnostic Test: Cy-TB test; Diagnostic Test: STANDARD F TB-Feron FIA test
- QuantiFERON-TB Gold Plus assay (Active Comparator): The QuantiFERON-TB Gold Plus assay will be used as the study's reference standard
  Interventions: Diagnostic Test: Cy-TB test; Diagnostic Test: STANDARD F TB-Feron FIA test

INTERVENTIONS:
Diagnostic Test: Cy-TB test — The study will include people with confirmed TB infection and negative controls to compare the specificity and sensitivity of the Cy-TB and TB-Feron tests versus the QFT-Plus assay
  Other Names: C-TB
Diagnostic Test: STANDARD F TB-Feron FIA test — The study will include people with confirmed TB infection and negative controls to compare the specificity and sensitivity of the Cy-TB and TB-Feron tests versus the QFT-Plus assay
  Other Names: TB-Feron

SUMMARY:
Introduction: The large reservoir of tuberculosis infections is a key driver of sustained tuberculosis (TB) incidence. Accurate diagnostic tests are crucial to correctly identify and treat people with TB infection, which is vital to eliminate TB globally. The Cy-TB skin test and STANDARD F TB-Feron FIA (TB-Feron) fluorescent immunoassay are two newly developed TB infection tests, which could offer quality and cost advantages over other commercially available TB infection tests, especially the standard TST test. Both tests have a higher sensitivity and specificity than the currently most used tuberculin skin test. The proposed study aims to evaluate the performance of these two tests for the diagnosis of TB infection, compared with the QuantiFERON-TB Gold Plus (QFT-Plus) assay.

Methods and analysis: This diagnostic accuracy study will employ a cross-sectional, observational design that aims to assess the accuracy of the Cy-TB and TB-Feron tests for diagnosing TB infection, using the QFT-Plus assay as the reference standard. The sensitivity and specificity will be reported. Three different cohorts of study participants will be recruited: Adults with microbiologically-confirmed pulmonary TB (n=100); Household contacts* of people with TB (n=200) and negative controls** (n=50). All participants will be examined with Cy-TB, TB-Feron, and QFT-Plus.

*Household contacts: of a person with TB are defined as members who live under the same roof as the person with pulmonary tuberculosis (PTB) or who meet the following conditions:

* Sleeping under the same roof or sharing a kitchen space as PTB-affected persons at least one night/week for three months before the person was diagnosed with PTB
* Staying under the same roof with PTB-affected persons for at least one hour/day and continuously five days/week for three months before the person was diagnosed with PTB

  * Negative controls are defined as people with a negative QFT-Plus result in the past year and likely to have no or very low rates of TB exposure history.

DETAILED DESCRIPTION:
Latent TB infection, hereafter referred to as TB infection, continues to be a significant driver of the global TB burden. A recent re-estimation using mathematical modeling demonstrated that to end TB by 2050, at least one-quarter of the global population living with TB infection would require TB preventive therapy (TPT).

The Tuberculin Skin Test (TST) and Interferon-Gamma Release Assays (IGRA) are the two preferred diagnostic methods for detecting TB infection. TST utilizes Tuberculin PPD RT 23 intradermally, which is low-cost and can easily be performed in the field. TST is currently the most frequently used TB infection test in Vietnam. However, TST has a low sensitivity and specificity, particularly in people who have had the BCG vaccine or are immunocompromised. IGRAs are more costly and more technically complex, requiring blood to be processed within a limited time-frame in a laboratory. Neither method is ideal for the detection of TB infection during community TB screening and contact investigations. Therefore, there is a need for a simple, affordable, and accurate diagnostic test for TB infection, to scale up TPT in Vietnam and globally.

Cy-TB (Serum Institute of India Pvt. Ltd, Pune, India) is a Mycobacterium Tuberculosis (MTB) antigen-based skin test, representing a new class of skin tests that were recommended by the World Health Organization in 2022. Cy-TB's MTB-specific antigens (ESAT6 and CFP10) are injected intradermally and provide results after 48-72 hours, similar to TST. The literature indicates that Cy-TB has a similar sensitivity and specificity to QuantiFERON TB Gold Plus.

Simplified versions of IGRAs are emerging, including TB-Feron (SD BIOSENSOR, INC, Gyeonggi-do, Republic of Korea). TB-Feron testing requires less manual handling than other IGRAs and testing takes only 15 minutes to complete after the specimen has been incubated for 16-24 hours. A recent clinical trial comparing the sensitivity and specificity of the TB-Feron against QIAreach QuantiFERON-TB (QIAGEN, Venlo, The Netherlands) showed that the TB-Feron has high accuracy in TB infection diagnosis (the sensitivity was 88.89% and specificity was 92.5%). There are currently no published evaluations comparing the performance of Cy-TB and TB-Feron to QFT-Plus in the literature.

Therefore, this study aims to evaluate the sensitivity and specificity of the Cy-TB and TB-Feron testing for the diagnosis of TB infection.

Aims

1. Main objective To evaluate the accuracy of the Cy-TB and TB-Feron tests versus the QFT-Plus assay as TB infection diagnostic methods in Vietnam, a high TB burden setting.
2. Specific objectives Objective 1: To verify the sensitivity of the Cy-TB and TB-Feron tests for TB infection diagnosis among adults with microbiologically confirmed pulmonary TB using QFT-Plus as the reference standard.

Objective 2: To evaluate the specificity and sensitivity of the Cy-TB test and TB-Feron tests compared to the QFT-Plus assay for the diagnosis of TB infections.

ELIGIBILITY:
Inclusion Criteria:

* All participants:

  * Agree to remain in contact and provide updated information as necessary, and have no current plans to relocate outside the designated area for the duration of the study
  * Capable of providing signed informed consent and informed assent (as appropriate)
* Group 1:

  + Microbiologically-confirmed pulmonary TB (either drug-susceptible TB or drug-resistant TB) via Xpert MTB/RIF or Xpert MTB/RIF Ultra (Cepheid, Sunnyvale, California) and abnormal chest X-ray (CXR) result*

  *To reduce the false positive rate of molecular diagnostic assays for M. tuberculosis
* Group 2:

  + Household contacts without symptoms of active TB disease of people with microbiologically-confirmed, pulmonary TB who initiated treatment with residents in Ha Noi, Vietnam.
* Group 3:

  * Known past negative IGRA test results among those at low risk for TB infection
  * No known and/or reported history of contact or exposure to either TB disease or M. tuberculosis bacteria.

Exclusion Criteria:

* All participants:

  + Declines to provide informed consent to participate in the study
* Groups 2 &3:

  * Presumed TB disease with symptoms (cough, fever, night sweats, unintentional weight loss) and/or an abnormal CXR result suggestive of TB disease
  * Microbiologically - or clinically-confirmed TB disease in all forms or report having taken treatment for TB disease.
  * History of TB infection (self-record or documented).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity | From study entry at the time of blood collection and Cy-TB injection until 72 hours post-injection, reported at the end of the trial.
  Point estimates of sensitivity with 95% confidence interval for the Cy-TB and TB-Feron tests, using the QFT-Plus assay as the reference standard

SECONDARY OUTCOMES:
Specificity | From study entry at the time of blood collection and Cy-TB injection until 72 hours post-injection, reported at the end of the trial.
  Point estimates of specificity with 95% confidence intervals of the Cy-TB and TB-Feron tests, using the QFT-Plus assay as the reference standard

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Lung Hospital, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nguyen HT, Vo LNQ, Codlin A, Forse R, Wingfield T, Sidney K, MacLean EL, Creswell J, Kirubi B, Davies Forsman L. Study protocol: diagnostic accuracy study comparing Cy-Tb and STANDARD F TB-Feron FIA tests for tuberculosis infection diagnosis in Vietnam. BMJ Open. 2024 Aug 9;14(8):e085614. doi: 10.1136/bmjopen-2024-085614. PMID 39122402